CLINICAL TRIAL: NCT04472390
Title: Study of Tapering and Discontinuing Biological DMARDs in Rheumatoid Arthritis Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201911037RIND
Record Dates: First submitted 2020-07-08; First posted 2020-07-15 (Actual); Last update posted 2020-07-15 (Actual); Status verified 2019-12

CONDITIONS: Rheumatoid Arthritis
Keywords: biological DMARDs
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Tapering: TNF-α inhibitors
- Discontinuing: TNF-α inhibitors

SUMMARY:
This study aims to analyses time to disease relapse of RA patients if TNF-α inhibitors are being tapered, the predictive factors that are associated with successful taper of TNF-α inhibitors. Also, investigate the effects associated with dose tapering of TNF-α inhibitors.

ELIGIBILITY:
Inclusion criteria:

Diagnosed of RA based on the 1987 American College of Rheumatology (ACR) criteria and/or 2010 ACR/EULAR classification criteria of RA depending on the time of diagnosis Age ≥ 20 years old TNF-α inhibitors was prescribed for RA patients refractory to csDMARDs (defined as csDMARD therapy for over 6 months) during 2003/5/2 - 2017/4/30 Dose reduction or discontinuation use of TNF-α inhibitors (2011/1/1-2019/4/30)

Exclusion criteria:

TNF-α inhibitors were discontinued or tapered due to adverse events such as infection, liver transaminase elevation, malignancy and neutropenia.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: There are 90 patients included in this cohort study, 89 patients underwent tapering of TNF-α inhibitors.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2019-12-03 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
time to disease relapse | hrough study completion, an average of 10 year
  me to relapse after tapering or discontinuing TNF-α inhibitors

CONTACTS AND LOCATIONS:
Overall Officials: Yen-Hui Chen, Principal Investigator — NTU Clinical Pharmacy School
Locations (1):
- National Taiwan University Hospital, Taipei, Zhongzheng District, Taiwan